CLINICAL TRIAL: NCT07145853
Title: "The Effect of Mandala Activity on Anxiety, Fatigue and Sleep Quality of Elderly Individuals Staying in a Nursing Home"
Brief Title: Mandala for Anxiety, Fatigue, and Sleep
Acronym: MANDALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Can Lafci, Lecturer, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MarmaraU-HB-CL-34
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Elderly Persons
Keywords: art therapy; Nursing Homes; Anxiety; fatigue; Sleep Quality
MeSH Terms: conditions — Anxiety Disorders; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Individuals included in the study will be randomized from the random.org website.
  Data will be collected twice in the intervention and control groups as pre-test and post-test. The pre-test of the study will be administered between May 2025-Septemb2025 and the post-test will be administered to individuals who completed the 8-week mandala activity in the intervention group. The descriptive questionnaire (Appendix-1) will not be applied in the post-test since the variables to be applied in the pre-test are fixed. Mandala activity will be applied to the intervention group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala activity group (Experimental): The application will last for 1-2 hours once a week for a total of 8 weeks.
  For individuals aged 65 years and over who meet the inclusion criteria and are included in the intervention group, a mandala draft in A4 format (21.0 cm x 29.7 cm) consisting of 8 round patterns to be determined in advance, and a dry paint set consisting of 12 colors for ease of use will be used. Quality dry paint will be used to prevent allergies
  Interventions: Other: Mandala activity
- Control Group (No Intervention): No intervention will be applied to the control group. The dry paint and mandala drafts necessary to overcome the deprivation of the control group will be left for them to do the activity after the study is completed.

INTERVENTIONS:
Other: Mandala activity — The application will last for 1-2 hours once a week for a total of 8 weeks.
  For individuals aged 65 years and over who meet the inclusion criteria and are included in the intervention group, a mandala draft in A4 format (21.0 cm x 29.7 cm) consisting of 8 round patterns to be determined in advance, and a dry paint set consisting of 12 colors for ease of use will be used. Quality dry paint will be used to prevent allergies
  Arms: Mandala activity group

SUMMARY:
Looking at the studies on social activity programs in individuals living in nursing homes in the literature, it was seen that the studies on Mandala therapy were limited. In this study, it is aimed to examine the effect of Mandala application, known as art therapy, on anxiety, fatigue and sleep quality in individuals living in nursing homes.

DETAILED DESCRIPTION:
In the world and in our country, the elderly population is increasing day by day. The average human life span is increasing as a result of the decrease in newborn rates, early diagnosis and treatment of chronic diseases due to developments in the field of medicine and technology, prevention of infectious diseases, increase in welfare level, increase in the level of education and health literacy of the society. The United Nations World Population Prospects 2022 report predicts that the number of individuals aged 65 and over will increase from 10% in 2022 to 16% in 2050. In Turkey, according to the Turkish Statistical Institute Statistics on the Elderly 2022 data, the proportion of the elderly population in the total population increased from 8.5% in 2017 to 9.9% in 2022. According to population projections, TÜİK predicts that the proportion of elderly population in Turkey will increase to 12.9% in 2030 and 16.3% in 2040.

Due to the increase in the elderly population, the care of the elderly population comes to the forefront as an important public health problem. With old age, which is an inevitable process, physiological, psychological, economic and social changes occur in individuals and adaptation problems are observed in individuals. Health care services of the elderly population is an important situation that requires a wide range of approaches. With old age, which is the last stage of life, there is a decrease in physical abilities, cognitive functions and activities of daily living. The elderly individual becomes more dependent on the environment as time passes. Due to the physiological changes brought about by old age, the risk of developing diseases increases. Many systems such as cardiovascular system, musculoskeletal system, gastrointestinal system, neuro-psychiatric system are affected in the elderly. Disability and disability increase in elderly individuals and therefore their quality of life deteriorates due to inadequacies in performing daily life activities.

Chronic diseases that occur due to aging make it more difficult for individuals to provide care for themselves. Care services for the elderly in need of care are provided formally and informally. Formal care is a set of professional care services provided by public/private institutions and organizations, while informal care is voluntary care provided by family, close relatives, neighbors or friends. In recent years, social changes due to many factors such as industrialization, modernization and urbanization affect the position of the elderly in society. Migrations from rural to urban areas, shrinking houses and increase in the rate of nuclear family, economic problems, increase in the employment rate of women, etc. Many factors cause problems in home care for the elderly. Elderly individuals who cannot find a place for themselves in the nuclear family may have to live alone or settle in public/private institutions or organizations such as nursing homes and move away from the environment and people they are used to.

Failure to address the psychological and social aspects holistically due to more emphasis on physical care in formal care leads to deterioration of cognitive functions in elderly individuals and difficulty in performing daily living activities. In addition, elderly people who are placed in institutions such as nursing homes may experience feelings such as isolation and feeling worthless due to the change in the environment and people who determine self-acceptance and respect. In old age, deterioration of the social support system consisting of spouse, family and friends, all kinds of losses, indifference, accepting old age as the last stage of life and additional diseases negatively affect psychological health. For these reasons, many psychological problems such as depression, anxiety, dementia, delirium and insomnia can be seen in the elderly. Social support is very important in coping with these problems.

Anxiety, fatigue and sleep quality are among the most important reasons that impair the functionality of elderly individuals and reduce their quality of life. It has been reported that living alone is an important risk factor for depression and suicide. This effect of living alone can be overcome with a social support system. Considering the prevalence of anxiety disorders in old age, it has been reported that the prevalence is between 14.2-29.4%. In a study conducted by Kırmızıoğlu et al. (2009) on elderly individuals in our country, general anxiety disorder was found to be 6.9% in this group.Risk factors associated with anxiety disorders include being female, being single, low education level, negative life events, comorbidities and childhood traumas.

In addition to physical, physiological and mental processes with aging, individuals' sleep quality and fatigue levels are affected as a result of lifestyle changes in the nursing home. In the systematic review study of Doris et al. it was reported that 27-50% of the elderly experienced moderate or severe fatigue. Sleep problems are increasing due to the aging process, and elderly individuals experience many conditions such as sleep quality, duration, continuity, and delay in sleep onset. The prevalence of sleep disorders in elderly individuals varies between 41.9% and 77%.

Nursing homes play a key role in the management of symptoms such as anxiety, fatigue and sleep quality in the elderly when social support cannot be provided by family and friends. This key role is made possible by providing social activity programs, meeting their psychological needs and housing in a healthy environment. In order for individuals living in nursing homes to participate more actively in life; work-oriented activities (handicraft, gardening, painting, wood painting), food activities (cooking, birthdays, tea time, etc.), exercise, cognitive therapies (cognitive stimulation therapies, reminiscence, etc.), music therapy, outdoor activities, prayer therapy and computer-aided activities can be done. These activity programs applied to the elderly improve the quality of life of the elderly. Cost-effective, therapeutic, non-pharmacological nursing interventions are needed to improve the quality of life of elderly individuals staying in nursing homes. Mandala is a Sanskrit term meaning circle or center, originating in India. Mandala is usually in the shape of a circle or square and is a painting method that allows transferring emotions and thoughts to paper. This activity is a colorful activity that can lead to problem solving. 'Manda' means energy or essence and 'La' means container. Mandala means a round container that holds or stores energy.Drawing a mandala starts by identifying a center point. There is always a human in the center. The picture or image created by the mandala is a reflection of the individual's current mood and self. Mandala painting is a psychotherapy technique that provides psychological support and healing.

Looking at the studies on social activity programs in individuals living in nursing homes in the literature, it was seen that the studies on Mandala therapy were limited. In this study, it is aimed to examine the effect of Mandala application, known as art therapy, on anxiety, fatigue and sleep quality in individuals living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* • Individuals aged 65 years and older with a score of 24 and above on the Mini Mental State Examination

  * Ability to use/hold a pen
  * Individuals without allergies,

Exclusion Criteria:

* Unable to communicate verbally
* Unable to act independently,
* Severe vision loss,
* People with neurological diseases such as stroke, Parkinson's, multiple sclerosis, dementia, etc,
* Has undergone any operation in the last six months,
* Individuals aged 65 and over diagnosed with cancer

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Score Measured by the Geriatric Anxiety Scale (GAS) [Score Range: 0-75] | Baseline and 8 weeks
  Anxiety will be assessed using the Geriatric Anxiety Scale (GAS). The scale consists of 23 items scored from 0 to 3, with a total score ranging from 0 to 75. Higher scores indicate higher levels of anxiety.

SECONDARY OUTCOMES:
Change in Fatigue Severity Measured by the Fatigue Severity Scale (FSS) [Score Range: 9-63] | Baseline and 8 weeks
  Fatigue will be assessed using the Fatigue Severity Scale (FSS), a 9-item self-report measure rated from 1 to 7. Total scores range from 9 to 63, with higher scores representing more severe fatigue.

OTHER OUTCOMES:
Change in Sleep Quality Score Measured by the Pittsburgh Sleep Quality Index (PSQI) [Score Range: 0-21] | Baseline and 8 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The instrument evaluates seven components of sleep quality, yielding a global score ranging from 0 to 21. A score greater than 5 indicates poor sleep quality. Higher scores reflect worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Can LAFÇI, PhDc, Principal Investigator — Marmara University
Locations (1):
- Faculty of Health Sciences, Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
"IPD will not be shared because of ethical and privacy considerations related to the vulnerable elderly population residing in a nursing home."